CLINICAL TRIAL: NCT04811326
Title: Latanoprost Plus NB-UVB Versus Each Alone in Non-segmental Vitiligo: Clinical and Laboratory Evaluation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shaimaa Fawzy Abdel-rady Abdel-latif (Other)
Responsible Party: Sponsor-Investigator, Shaimaa Fawzy Abdel-rady Abdel-latif, investigator, Aswan University Hospital
Organization: Aswan University Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 504/1/21
Record Dates: First submitted 2021-03-07; First posted 2021-03-23 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Non-segmental Vitiligo
MeSH Terms: interventions — Latanoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NB-UVB radiation (Active Comparator): will expose to 2 sessions/week of NB-UVB radiation, for 3 months.
  Interventions: Radiation: NB-UVB
- Latanoprost (Active Comparator): latanoprost 0.005%, will be applied after microneedling, by using 1.5-2 mm needle length dermapen, of vitiligenous patches. The procedure will be repeated once weekly for 3 months (12 sessions).
  Interventions: Drug: Latanoprost
- latanoprost + NB-UVB (Active Comparator): (latanoprost + NB-UVB group): latanoprost 0.005%, will be applied after microneedling of vitiligenous patches in the same day of NB-UVB sessions in the same manner of group 2.
  Interventions: Radiation: NB-UVB; Drug: Latanoprost
- healthy individuals (No Intervention): healthy individuals as control group

INTERVENTIONS:
Radiation: NB-UVB — radiation
  Other Names: narrow band ultraviolet B
  Arms: NB-UVB radiation; latanoprost + NB-UVB
Drug: Latanoprost — eye drops
  Other Names: latanoprost eye drops
  Arms: Latanoprost; latanoprost + NB-UVB

SUMMARY:
The aim of the study is to evaluate the efficacy of different lines of therapies on the TWEAK serum level in patients with non-segmental vitiligo.

DETAILED DESCRIPTION:
the study is to evaluate the efficacy of NB-UVB, latanoprost, and combination of them on the TWEAK serum level in patients with non-segmental vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-segmental vitiligo of any age and gender.

Exclusion Criteria:

* History of vitiligo treatment with topical, systemic or biological agents prior to the study for at least 3 weeks.
* Pregnancy and lactation.
* Infections
* Patients with other autoimmune diseases.
* Patients with chronic diseases: cardiac diseases, hepatic disorders, hematologic disease, chronic renal failure or malignancies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2024-02-13 (Estimated); Study Completion 2024-03-13 (Estimated)

PRIMARY OUTCOMES:
serum TWEAK in vitiligo | 3months
  measurement of serum Tumor necrosis factor weak inducer of apoptosis (TWEAK)"pg/ml"; in vitiligo patients before and after treatment with NB-UVB, Latanoprost and their combination, all in comparison with healthy individuals, using ELISA (enzyme-linked immunosorbent assay)

SECONDARY OUTCOMES:
treatment of vitiligo | 3 months
  clinical evaluation: Assessment of the disease severity in non-segmental vitiligo will be performed by using vitiligo area severity index (VASI score) before and after treatment with NB-UVB, latanoprost application applied after microneedling, by using 1.5-2 mm needle length dermapen, of vitiligenous patches, or combination of both of them. Patients will be photographed at baseline and after 3 months of regular treatment by using high resolution digital camera conon EOS 1300D 18 megapixels (made in Taiwan), photography will be done in standard light and distance.

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa A El Taieb, prof., Study Chair — Prof. and Head of Dermatology, Venereology and Andrology department, Aswan University, Egypt
Locations (1):
- faculty of medicine, Aswan University, Aswān, Aswan Governorate, Egypt